CLINICAL TRIAL: NCT02735850
Title: A Randomized Phase II Trial of the Combination of SBRT With L19-IL2 in Patients With Limited Metastatic Non-small Cell Lung Cancer (NSCLC)
Brief Title: Combination of SABR and L19-IL2 in Patients With Stage IV Lung Cancer (ImmunoSABR)
Acronym: ImmunoSABR
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Not yet submitted, unclear timelines
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other); Karolinska Institutet (Other); University of Oxford (Other); KU Leuven (Other); Copenhagen University Hospital at Herlev (Other); Catholic University of the Sacred Heart (Other); The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Oligometa's L19-IL2
Record Dates: First submitted 2016-03-22; First posted 2016-04-13 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2016-04

CONDITIONS: NSCLC Stage IV; Limited Metastatic Disease
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — L19-IL2 immunocytokine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ablative SBRT to all (max 3) sites followed by L19-IL2 (Experimental): Ablative cohort
  Interventions: Drug: L19-IL2; Radiation: SBRT
- Ablative SBRT to all (max 3) sites (Active Comparator): Ablative cohort
  Interventions: Radiation: SBRT
- SBRT 1 site, L19-IL2 and then standard of care (Experimental): Non-ablative cohort
  Interventions: Radiation: SBRT
- Standard of care (Active Comparator): Non-ablative cohort
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: L19-IL2 — L19-IL2 added to SBRT
  Arms: Ablative SBRT to all (max 3) sites followed by L19-IL2
Radiation: SBRT
  Arms: Ablative SBRT to all (max 3) sites; Ablative SBRT to all (max 3) sites followed by L19-IL2; SBRT 1 site, L19-IL2 and then standard of care
Other: No intervention
  Arms: Standard of care

SUMMARY:
This will be a phase II trial testing if the combination of SBRT and L19-IL2 improves the progression free survival in patients with limited metastatic non-small cell lung cancer (NSCLC). Treatment will be divided in two cohorts: patients eligible for ablative stereotactic body radiotherapy to all metastatic sites (treatment with curative intent) and patients not eligible for stereotactic body radiotherapy to all sites (life prolongation).

DETAILED DESCRIPTION:
IMMUNOSABR will include 138 patients. The trialpopulation will be divided in two cohorts: patients eligible for ablative stereotactic body radiotherapy to all metastatic sites (treatment with curative intent) and patients not eligible for stereotactic body radiotherapy to all sites (life prolongation).In this single stage phase II trial we aim to demonstrate absolute increase in progression free survival at two years. . PFS will be determined as the time between randomization and disease progression, according to RECIST 1.1, death due to any cause or last patient contact alive and progression-free. Patients will be randomized between control (no L19-IL2) and experimental arms (with L19-IL2) in a 1:1 ratio. The accrual period will be 29 months (or 2.41 years) and the minimum follow-up will be 24 months (or 2 years), making the total study duration 53 months (or 4.41 years). Comparison between control and experimental arms will be done using the Log-Rank statistic. This test for superiority will be one-sided with a desired type I error of 0.10 and power of 0.80. The randomization allocation is 1:1.

Primary endpoint and power calculation For the ablative cohort: the expected 2-year PFS is 20% in the control arm (arm A) and 40% in the experimental arm ( arm B). The study is therefore powered to test for a difference in PFS at 2 years of 20%. The null hypothesis (H0) is that there is no difference in PFS between arm A and arm B. This results in a sample size of 72 patients evenly divided over two arms with 36 patient per arm. Considering a dropout rate of 10% from current experience, the actual amount of patients will be 40 per arm or 80 in total.

For the non-ablative cohort: the expected 2-year PFS is 10% in the control arm (arm C) and 30% in the experimental arm (arm D) The study is therefore powered to test for a difference in PFS at 2 years of 20%. The null hypothesis (H0) is that there is no difference in PFS between arm C and arm D. This resuls in a sample size of 52 patients evenly divided over two arms with 26 patient per arm. Considering a dropout rate of 10% from current experience, the actual amount of patients will be 29 per arm or 58 in total.

The total number of patients needed for the trial is the sum of the amount of patients in the ablative cohort (80 patients) and the amount of patients in the non-ablative cohort (58 patients): 138 patients.

Secondary endpoints Simple univariate comparisons of outcome and toxicity will be made between both treatment arms in each cohort using Chi-square tests for categorical data and independent samples t-tests for scale data. Secondary study parameter(s): Overall survival (OS) will be assessed using survival tables and Kaplan-Meier curves. OS will be calculated from the day of randomisation. Abscopal response, which can only be measured in the non-ablative cohort (with at least one non-irradiated target lesion) will measured as best response between experimental and standard treatment arms. Quality of life (EORTC QLQ-C30 version 3.0 and QLQ-LC13 questionnaires) will be recorded at regular intervals. Average changes in quality of life will be reported in terms of absolute differences in scores, and also in terms of minimally clinically relevant changes.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed limited metastatic NSCLC patients. Two cohorts of patients are allowed:

  * Synchronous oligometastatic eligible for ablative stereotactic body radiotherapy to all sites. These patients will have a maximum of 3 metastatic lesions (excluding the brain) eligible for ablative treatment using SABR.,
  * Other oligometastatic patients with up to 10 metastatic lesions, not eligible for ablative stereotactic body radiotherapy, that have controlled disease (i.e. no progressive disease according to RECIST 1.1) following primary chemotherapy with a platinum doublet, with at least one measurable lesion that is not subjected to stereotactic body radiotherapy (SABR),.
* Radiological images documenting this lesion should be no older than 28 days before study enrolment.
* Age of 18 y or older.
* Prior treatments are allowed but must be discontinued for at least 4 weeks before enrolment.
* All radiology studies must be performed within 28 days prior to registration
* WHO performance status 0-2;
* Adequate bone marrow: Normal white blood cell count and formula, normal platelet count, no anemia requiring blood transfusion or erythropoietin;
* Adequate hepatic function: total bilirubin ≤ 1.5 x upper limit of normal (ULN) for the institution; ALT, AST, and alkaline phosphatase ≤ 2.5 x ULN for the institution or <= 5 in case of liver metastasis);
* Adequate renal function: creatinine clearance at least 60 ml/min;
* The patient is capable of complying with study procedures;
* Life expectancy of at least 12 weeks;
* Men and women with reproductive potential must be willing to practice acceptable methods of birth control during the study and for up to 12 weeks after the last dose of study medication.
* Signed and dated written informed consent;

Exclusion Criteria:

* NSCLC with activating ALK/EGFR of ROS mutations.
* SABR required to brain metastasis
* Previous chemotherapy other than a platinum doublet.
* Patients with progressive disease following initial chemotherapy.
* Previous chemotherapy for more than 25 weeks.
* Previous radiotherapy to an area that would be re-treated by SABR;
* Other active malignancy or malignancy within the last 2 years (with exception of localized skin basal/squamous cell carcinoma, bladder in situ carcinoma);
* History of allergy to intravenously administered proteins/peptides/antibodies;
* HIV infection, active infection, or active hepatitis;
* Chronic systemic use of corticosteroids used in the management of cancer or non-cancer-related illness;
* Acute or sub-acute coronary syndromes within the last year, acute inflammatory heart disease, heart insufficiency or irreversible cardiac arrhythmias;
* Impaired cardiac function defined as left ventricular ejection fraction (LVEF) < 50 % (or below the study site's lower limit of normal) as measured by MUGA or ECHO. (LVEF measurements dating back up to 8 weeks will be acceptable in the absence of intercurrent use of potentially cardiotoxic treatment or cardiac medical history).
* Uncontrolled hypertensive disease
* History or evidence of active autoimmune disease;
* Severe diabetic retinopathy (neoangiogenesis targeted by L19 outside the tumor)
* Major trauma, including surgery, within 4 weeks prior to entering the study (neoangiogenesis targeted by L19 outside the tumor)
* Any underlying medical or psychiatric condition which in the opinion of the investigator will make administration of study drug hazardous or hinder the interpretation of study results (e.g., AE);
* Unstable or serious concurrent uncontrolled medical conditions;
* Pregnancy or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Improved progression free survival | 2 years after treatment
  Test the combination of SBRT and L19-IL2 in progression free survival (follow-up visit)

SECONDARY OUTCOMES:
Overall survival | 2 years after treatment
  Follow-up visit
Quality of life | 2 years after treatment
  Questionnaire
Abscopal responses defined as partial or complete remission to RECIST 1.1 of lesions outside the radiotherapy field (only possible in the non-ablative cohort) | 20 weeks (during treatment)
  Scan
Associative biomarkers | 20 weeks (during treatment)
  Blood withdrawal. ED-B of fibronectin (periferal blood), changes in the different fractions of periferal blood, mononuclear cells like cytotoxic T-cells, NK cells, memory T-cells (periferal blood), inflammatory cytokines (periferal blood). ED-B expression in the tumor (biopsies), HLA class I expression (tumor biopsies).
Determination of hypoxia status by [18F]HX4-Positron Emmission Tomography (PET) (optional) | 20 weeks (during treatment)
  Scan

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, MD, PhD, Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- MAASTRO clinic, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided